CLINICAL TRIAL: NCT03696004
Title: Outcome of Neo-adjuvant Chemotherapy Followed by Breast Conservative Surgery in Breast Cancer in Upper Egypt
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Sammani Ali Muhammad, General Surgery Resident, Assiut University
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SAMuhammad
Record Dates: First submitted 2018-10-03; First posted 2018-10-04 (Actual); Last update posted 2018-10-04 (Actual); Status verified 2018-05

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Retros FEC-100 +BRS (Active Comparator): Contains record of already treated patients with six cycles of FEC-100 Fluorouracil ,Epirubicin and Cyclophosphamide and later had Breast conservative Surgery(BRS)
  Interventions: Drug: FEC-100
- PROS 30 FEC-100 +BRS (Active Comparator): These are new patients who will be treated with six cycles of FEC-100 (Flourouracil,Epirubicin and Cyclophosphamide) and will undergo Breast Conservative Surgery (BRS)after 6 weeks
  Interventions: Drug: FEC-100

INTERVENTIONS:
Drug: FEC-100 — Patients will recieve six cycles of FEC-100 and Breast conservative surgery after 4-6 weeks
  Other Names: Breast Conservative Surgery

SUMMARY:
Systemic chemotherapy along with radiotherapy has been successfully used to post-operatively manage patients following tumour resection in breast cancer.

This was further supported with clinical trials conducted in the 1970s and 1980s which shows significant improvement in progression-free of tumours and overall survival rates in patients who undergo chemotherapy for operable breast cancer.(1)-(2) Neoadjuvant chemotherapy on the other hand, involves the administration of the chemotherapeutic agents some weeks before appropriate breast surgery. This induces reduction in the tumour size and allows for breast conservative surgery instead of mastectomy in some cases.

Techniques for tumour localization in neoadjuvant chemotherapy using metallic markers allowing lower excision of breast tissue without compromising margins and breast conservation being feasible in many patients have evolved over time.(3)-(7)-(9) However, there are recent concerns questioning the increase use of neoadjuvant chemotherapy in breast cancer it as it may not be beneficial to patients in the long run.(10)

DETAILED DESCRIPTION:
This will consist of six cycles of FEC-100 regimen followed by surgery. The decision on the type of surgery (breast conservative surgery or mastectomy) will be taken on the final assessment of the disease after the six cycle.

Neoadjuvant chemotherapy regimen will consist of six cycles of fluorouracil 500mg/m2 , epirubicin 75mg/m2 and cyclophosphamide 500mg/m2 administered intravenously at three week interval.

Surgery was planned to be performed within 4-6 weeks after the six course of chemotherapy.

ELIGIBILITY:
Inclusion Criteria:1- female patients diagnosed with breast cancer and are attending oncology or surgical unit of Assiut university hospital .

2- breast cancer will be diagnosed by core-needle biopsy. 3- all patients must have complete history and physical examination (including careful assessment of breast and axillary lymph nodes).

4- All patients must have routine laboratory tests (CBC, liver and renal function tests, and alkaline phosphatase) and radiological tests (chest x-ray, pelvic-abdominal ultrasound, bilateral mammography with confirmatory ultrasound and complete echocardiography to assess the cardiac function).

5- written consent from patients.

-

Exclusion Criteria:

* 1- Elderly patients more than 70years old. 2- Previous treatment for breast cancer. 3- Presence of co-existing malignancies. 4- Pregnancy or lactation at time of diagnosis. 5- Severe renal, hepatic or haematological abnormalities. 6- Bilateral breast cancer. 7- advanced breast cancer

Ages: 18 Years to 69 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Female patients diagnosed with breast cancer
Enrollment: 45 (Estimated)
Dates: Start 2018-12 (Estimated); Primary Completion 2019-06 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
Tumour size measurement | 18 WEEKS
  Measurement of tumuor size before and after six courses of FEC-100

CONTACTS AND LOCATIONS:
Overall Officials: Hisham A Riad, PhD, Study Chair — Assiut University; Samir S Mohamed, PhD, Study Director — Assiut University
Locations (1):
- Assiut University Hospital, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Espinosa-Bravo M, Sao Aviles A, Esgueva A, Cordoba O, Rodriguez J, Cortadellas T, Mendoza C, Salvador R, Xercavins J, Rubio IT. Breast conservative surgery after neoadjuvant chemotherapy in breast cancer patients: comparison of two tumor localization methods. Eur J Surg Oncol. 2011 Dec;37(12):1038-43. doi: 10.1016/j.ejso.2011.08.136. Epub 2011 Sep 21. PMID 21940138
- [Background] Bobin JY, Al-Khaledi K, Ahmad J. Breast conservative surgery for operable invasive ductal carcinoma after neoadjuvant chemotherapy or hormonal therapy- a challenge for breast surgeon: a review based on literature and experience. Gulf J Oncolog. 2011 Jan;(9):45-51. PMID 21177208
- [Background] Schwartz GF, Meltzer AJ, Lucarelli EA, Cantor JP, Curcillo PG 2nd. Breast conservation after neoadjuvant chemotherapy for stage II carcinoma of the breast. J Am Coll Surg. 2005 Sep;201(3):327-34. doi: 10.1016/j.jamcollsurg.2005.03.015. PMID 16125064
- [Background] Van Praagh I, Cure H, Leduc B, Charrier S, Le Bouedec G, Achard JL, Ferriere JP, Feillel V, De Latour M, Dauplat J, Chollet P. Efficacy of a primary chemotherapy regimen combining vinorelbine, epirubicin, and methotrexate (VEM) as neoadjuvant treatment in 89 patients with operable breast cancer. Oncologist. 2002;7(5):418-23. doi: 10.1634/theoncologist.7-5-418. PMID 12401904
- [Background] Kuerer HM, Singletary SE, Buzdar AU, Ames FC, Valero V, Buchholz TA, Ross MI, Pusztai L, Hortobagyi GN, Hunt KK. Surgical conservation planning after neoadjuvant chemotherapy for stage II and operable stage III breast carcinoma. Am J Surg. 2001 Dec;182(6):601-8. doi: 10.1016/s0002-9610(01)00793-0. PMID 11839324
- [Background] Vaidya JS, Massarut S, Vaidya HJ, Alexander EC, Richards T, Caris JA, Sirohi B, Tobias JS. Rethinking neoadjuvant chemotherapy for breast cancer. BMJ. 2018 Jan 11;360:j5913. doi: 10.1136/bmj.j5913. No abstract available. PMID 29326104
- [Result] Abdel-Bary N, El-Kased A, Aiad H. Does neoadjuvant chemotherapy increase breast conservation in operable breast cancer: an Egyptian experience. Ecancermedicalscience. 2009;3:104. doi: 10.3332/ecancer.2008.104. Epub 2009 Apr 9. PMID 22275993
- [Result] Inaji H, Komoike Y, Motomura K, Kasugai T, Sawai Y, Koizumi M, Nose T, Koyama H. Breast-conserving treatment after neoadjuvant chemotherapy in large breast cancer. Breast Cancer. 2002;9(1):20-5. doi: 10.1007/BF02967542. PMID 12196717